CLINICAL TRIAL: NCT03166124
Title: Pharmacokinetics and Glucodynamics of LY900014 Compared to Insulin Lispro Following Single Dose Administration in Elderly and Younger Adults With Type 1 Diabetes Mellitus
Brief Title: A Study of LY900014 in Elderly and Younger Adult Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16637; I8B-MC-ITRR (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Elderly Adults LY900014 (Experimental): Single, subcutaneous (SC) 15-U dose of LY900014 in the elderly adult group.
  Interventions: Drug: LY900014
- Elderly Adults Insulin Lispro (Active Comparator): Single, SC 15-U dose of insulin lispro (Humalog) in in the elderly adult group.
  Interventions: Drug: Insulin Lispro
- Younger Adults LY900014 (Experimental): Single, SC 15-U dose of LY900014 in the younger adult group.
  Interventions: Drug: LY900014
- Younger Adults Insulin Lispro (Active Comparator): Single, SC 15-U dose of insulin lispro (Humalog) in the younger adult group.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: Elderly Adults LY900014; Younger Adults LY900014
Drug: Insulin Lispro — Administered SC
  Other Names: Humalog; LY275585
  Arms: Elderly Adults Insulin Lispro; Younger Adults Insulin Lispro

SUMMARY:
The purpose of this study is to compare LY900014 with insulin lispro (Humalog) in elderly and younger adults with type 1 diabetes mellitus.

Screening is required within 28 days prior to the start of the study. For each participant, the total duration of the clinical trial will be between 3 to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female participants with Type 1 Diabetes Mellitus (T1DM)
* Have a body mass index (BMI) of 18.5 to 30.0 kilogram per meter square (kg/m²)
* Have a glycated hemoglobin (HbA1c) less than (<)9.0 percent (%)
* Have had no episodes of severe hypoglycaemia in the last 6 months

Exclusion Criteria:

* Have a history or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (apart from T1DM), hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data
* Have a history of renal impairment
* Have a history of deep vein thrombosis of the leg or repeated episodes of deep leg vein thrombosis in first-degree relatives
* Have proliferative retinopathy or maculopathy and/or severe neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-11-18 (Actual); Study Completion 2017-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Neuss

REFERENCES:
- [Derived] Leohr J, Dellva MA, Carter K, LaBell E, Linnebjerg H. Ultra Rapid Lispro (URLi) Accelerates Insulin Lispro Absorption and Insulin Action vs Humalog(R) Consistently Across Study Populations: A Pooled Analysis of Pharmacokinetic and Glucodynamic Data. Clin Pharmacokinet. 2021 Nov;60(11):1423-1434. doi: 10.1007/s40262-021-01030-0. Epub 2021 May 27. PMID 34041713
- [Derived] Linnebjerg H, Zhang Q, LaBell E, Dellva MA, Coutant DE, Hovelmann U, Plum-Morschel L, Herbrand T, Leohr J. Pharmacokinetics and Glucodynamics of Ultra Rapid Lispro (URLi) versus Humalog(R) (Lispro) in Younger Adults and Elderly Patients with Type 1 Diabetes Mellitus: A Randomised Controlled Trial. Clin Pharmacokinet. 2020 Dec;59(12):1589-1599. doi: 10.1007/s40262-020-00903-0. PMID 32468447

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 2-period, crossover study, up to 10-hour euglycemic clamp in which participants were randomized to 1 of 2 treatment sequences: LY900014 in Period 1 switching to Humalog period 2 or Humalog in Period 1 switching to LY900014 in Period 2. A washout period of 3 to 15 days occurred between study drug administration.
Groups:
- Sequence 1 AB Elderly Adults: Sequence 1:
  A: Single, subcutaneous (SC) 15-U dose of LY900014 in Period 1. B: Single, SC 15-U dose of Humalog in Period 2. Washout period of 3-15 days between study drug administration.
- Sequence 1 AB Younger Adults: Sequence 1 A: Single, SC 15-U dose of LY900014 in Period 1. B: single, SC 15-U dose of Humalog in Period 2. Washout 3-15 days between study drug administration.
- Sequence 2 BA Elderly Adults: Sequence 2:
  B: Single, SC 15-U dose of Humalog in Period 1. A: Single, SC 15-U dose of LY900014 in Period 2. A Washout period of 3-15 days between study drug administration.
- Sequence 2 BA Younger Adults: Sequence 2:
  B: Single, SC 15-U dose of Humalog in Period 1. A: Single SC 15-U dose of LY900014 in Period 2. A Washout period of 3-15 days between study drug administration.
Period: Treatment Period 1
Arm/Group | Sequence 1 AB Elderly Adults | Sequence 1 AB Younger Adults | Sequence 2 BA Elderly Adults | Sequence 2 BA Younger Adults
Started | 20 | 20 | 19 | 21
Received at Least One Dose of Study Drug | 20 | 20 | 18 | 21
Completed | 20 | 20 | 18 | 21
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Wash-out Period
Arm/Group | Sequence 1 AB Elderly Adults | Sequence 1 AB Younger Adults | Sequence 2 BA Elderly Adults | Sequence 2 BA Younger Adults
Started | 20 | 20 | 18 | 21
Completed | 20 | 18 | 17 | 20
Not Completed | 0 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1 AB Elderly Adults | Sequence 1 AB Younger Adults | Sequence 2 BA Elderly Adults | Sequence 2 BA Younger Adults
Started | 20 | 18 | 17 | 20
Completed | 20 | 18 | 17 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Elderly Adults: Male and female participants age 65 or older inclusive.
- Younger Adults: Male and female participants age 18 to 45 inclusive.
- Total: Total of all reporting groups
Arm/Group | Elderly Adults | Younger Adults | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (2.7) | 32.0 (6.8) | 49.8 (19.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 22 | 28 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 39 | 41 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 39 | 41 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 39 | 41 | 80
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 76.66 (12.61) | 78.39 (10.00) | 77.55 (11.41)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Insulin Lispro Area Under the Concentration Versus Time Curve (AUC) for Each Treatment Arm
Description: Pharmacokinetics: Insulin lispro AUC from time zero to 10 hours postdose [AUC(0-10h)] for each treatment arm.
Time Frame: Day 1: Pre-dose, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, 300, 360, 420, 480, 540, and 600 minutes post-dose
Population: All participants who received at least one dose of study drug and have measurable insulin lispro concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole * hour per Liter (pmol*h/L)
Groups:
- Elderly Adults LY900014: All elderly adults who received a single 15-U SC dose LY900014.
- Elderly Adults Humalog: All elderly adults who received a single 15-U SC dose Humalog.
- Younger Adults LY900014: All younger adults who received a single 15-U SC dose LY900014.
- Younger Adults Humalog: All younger adults who received single 15-U SC dose Humalog.
Arm/Group | Elderly Adults LY900014 | Elderly Adults Humalog | Younger Adults LY900014 | Younger Adults Humalog
Number analyzed (Participants) | 37 | 37 | 40 | 39
picomole * hour per Liter (pmol*h/L) | 1430 (26) | 1400 (29) | 1210 (24) | 1170 (30)
Statistical Analysis 1: Comparison: Elderly Adults LY900014 vs Elderly Adults Humalog; Geometric LSMeans were controlled for injection site, study period, and sequence as fixed effects, and subject within sequence as a random effect; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric LSMeans = 1.02, 95% CI 2-sided [0.953 to 1.10]
Statistical Analysis 2: Comparison: Younger Adults LY900014 vs Younger Adults Humalog; Geometric Least Squares Means (LSMeans) were controlled for injection site, study period, and sequence as fixed effects, and subject within sequence as a random effect; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric LSMeans = 1.03, 95% CI 2-sided [0.974 to 1.09]

2. Secondary Outcome: Total Amount of Glucose Infused (Gtot) Over Duration of Clamp for Each Treatment Arm
Description: Glucodynamics: Gtot is the total glucose infusion over the clamp duration (10 hours) and is used to measure the study drug action over time as measured by the euglycemic clamp procedure.
Time Frame: Every minute starting from the pre-dose and throughout the duration of the clamp until 10 hours post-dose
Population: All participants who received at least one dose of study drug and completed at least one clamp procedure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram per kilogram (mg/kg)
Groups:
- Younger Adults Humalog: All younger adults who received a single 15-U SC dose Humalog.
Arm/Group | Elderly Adults LY900014 | Elderly Adults Humalog | Younger Adults LY900014 | Younger Adults Humalog
Number analyzed (Participants) | 37 | 35 | 40 | 39
milligram per kilogram (mg/kg) | 1140 (42) | 1090 (43) | 1170 (33) | 1150 (30)
Statistical Analysis 1: Comparison: Elderly Adults LY900014 vs Elderly Adults Humalog; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric LSMeans = 1.04, 95% CI 2-sided [0.96 to 1.12]
Statistical Analysis 2: Comparison: Younger Adults LY900014 vs Younger Adults Humalog; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric LSMeans = 1.02, 95% CI 2-sided [0.94 to 1.10]

ADVERSE EVENTS:
Time Frame: Baseline to end of study (up to 39 days)
Description: All participants who received at least one dose of study drug.
Groups:
- Elderly Adults LY900014: Single, subcutaneous (SC) 15-U dose of LY900014.
- Elderly Adults Humalog; Younger Adults Humalog: Single, SC 15-U dose of Humalog.
- Younger Adults LY900014: Single, SC 15-U dose of LY900014.
Arm/Group | Elderly Adults LY900014 | Elderly Adults Humalog | Younger Adults LY900014 | Younger Adults Humalog
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38 | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38 | 1/40 | 0/39
Other Adverse Events (participants affected / at risk) | 5/37 | 7/38 | 3/40 | 6/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elderly Adults LY900014 (N=37) | Elderly Adults Humalog (N=38) | Younger Adults LY900014 (N=40) | Younger Adults Humalog (N=39)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elderly Adults LY900014 (N=37) | Elderly Adults Humalog (N=38) | Younger Adults LY900014 (N=40) | Younger Adults Humalog (N=39)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (4) | 5 (5) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT03166124/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT03166124/SAP_001.pdf